CLINICAL TRIAL: NCT02664909
Title: Topical (Intra-Articular) Tranexamic Acid and Transfusion Rates Following Hip Hemiarthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-058SF-2; 0546934781 (Other: UCHC)
Record Dates: First submitted 2016-01-13; First posted 2016-01-27 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Femoral Neck Fractures
Keywords: Hip Hemiarthroplasty; Tranexamic Acid; Topical; Blood Transfusion
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Patients will receive 1 gram of topically applied tranexamic acid into their surgical wound at the time of wound closure during their hip hemiarthroplasty surgery. 1 gram of tranexamic acid will be mixed with normal saline to a total volume of 50 cc, half of which will be delivered intra-articularly and half of which will be delivered in the subfascial space.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Patients will receive 50 cc of topically applied normal saline into their surgical wound at the time of wound closure during their hip hemiarthroplasty surgery. Half of this 50 cc dose of normal saline will be delivered intra-articularly and half will be delivered in the subfascial space.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Drug: Placebo (saline)
  Arms: Placebo

SUMMARY:
This study is a double-blinded placebo-controlled clinical trial evaluating the efficacy of 1 gram of topically applied tranexamic acid vs. saline placebo for the reduction of transfusion following hip hemiarthroplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip hemiarthroplasty surgery for a displaced femoral neck fracture

Exclusion Criteria:

* History of hemophilia, history of deep vein thrombosis, history of pulmonary embolism, history of thrombophilia, history of chronic renal failure
* Patients with coronary ischemia (active or within the past calendar year), patients who have suffered a myocardial infarction, undergone percutaneous coronary intervention, undergone coronary artery bypass grafting, or undergone any revascularization procedure within the past calendar year
* Patients with active subarachnoid hemorrhage, acquired defective color vision, patients who sustained a pathologic fracture (fracture through a neoplastic lesion), or patients who are pregnant
* Patients with a known allergy to tranexamic acid
* Patients taking Warfarin, Dabigatran, Rivaroxaban, Apixaban, and Fresh Frozen Plasma

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- Tranexamic Acid: Patients will receive 1 gram of topically applied tranexamic acid into their surgical wound at the time of wound closure during their hip hemiarthroplasty surgery. 1 gram of tranexamic acid will be mixed with normal saline to a total volume of 50 cc, half of which will be delivered intra-articularly and half of which will be delivered in the subfascial space.
  Tranexamic Acid
- Placebo: Patients will receive 50 cc of topically applied normal saline into their surgical wound at the time of wound closure during their hip hemiarthroplasty surgery. Half of this 50 cc dose of normal saline will be delivered intra-articularly and half will be delivered in the subfascial space.
  Placebo (saline)
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 17 | 19
Completed | 15 | 16
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 83 (8.6) | 83 (9.6) | 83 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 17 | 19 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Needed Transfusions
Description: The rate of transfusion will be calculated for each study group.
Time Frame: From the time of surgery until 2-4 days post-operative (length of inpatient hospital stay)
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 17 | 19
Participants | 0 | 5

2. Secondary Outcome: Inpatient Transfusion Amount
Description: The transfusion amount will be calculated for each study group.
Time Frame: 2-4 days post-operative (length of inpatient hospital stay)
Measure: Mean (Standard Deviation); unit: unit of blood (250 cc)
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 17 | 19
unit of blood (250 cc) | NA (NA) — No patient received transfusions | 1.2 (0.45)

3. Secondary Outcome: Difference Between Pre/Post-operative Hemoglobin
Time Frame: Pre-operative hemoglobin level vs. post-operative day 1 hemoglobin level
Measure: Mean (95% Confidence Interval); unit: grams per deciliter
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 17 | 19
grams per deciliter | 1.45 [1.10 to 1.81] | 1.48 [0.71 to 2.25]

4. Secondary Outcome: Difference Between Pre/Post-operative Hematocrit
Time Frame: Pre-operative hematocrit level vs. post-operative day 1 hematocrit level
Measure: Mean (95% Confidence Interval); unit: percent of blood that is red blood cells
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 17 | 19
percent of blood that is red blood cells | 4.1 [2.98 to 5.17] | 4.4 [2.18 to 6.56]

5. Secondary Outcome: Length of Inpatient Hospital Stay
Time Frame: From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever comes first, assessed up to 42 days post-operatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 17 | 19
days | 3.9 (1.1) | 4.8 (1.9)

6. Secondary Outcome: Number of Participants With Post-operative Complications
Time Frame: Admission to second post-operative visit (4-6 weeks post-operative)
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 17 | 19
Participants | 6 | 11

7. Secondary Outcome: Inpatient Hospitalization Cost
Time Frame: Collected 4-6 weeks post-operative
Population: Data was not gathered for this outcome measure and therefore never analyzed.
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/19
Other Adverse Events (participants affected / at risk) | 6/17 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=17) | Placebo (N=19)
inpatient treatment for myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
demand ischemia (Cardiac disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=17) | Placebo (N=19)
1 readmission for a fall with a contralateral hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
altered mental state (Psychiatric disorders) | 0 (0) | 1 (1)
syncope (Cardiac disorders) | 0 (0) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 1 (1)
agitation (Psychiatric disorders) | 0 (0) | 2 (2)
urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
fever (General disorders) | 3 (3) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
foley catheter (Renal and urinary disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT02664909/Prot_SAP_000.pdf